CLINICAL TRIAL: NCT05168787
Title: Efficacy and Safety of Sacubitril/Valsartan in African American Patients With Heart Failure With Reduced Ejection Fraction
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 047.PHA.2020.A
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril belongs to a class of drugs called neprilysin inhibitors and valsartan belongs to a class of drugs called angiotensin receptor blockers (ARBs). They work by relaxing blood vessels so that blood can flow more easily, which makes it easier for your heart to pump blood to your body.

SUMMARY:
There is limited long-term evidence specific to AAs with HFrEF on sacubitril/valsartan therapy. Plasma NT-proBNP levels are lower in AA individuals as compared to Caucasian individuals in general. However, the mechanism of action of sacubitril specifically targets the activity of BNP. Therefore, there is the potential that the mechanism of action of sacubitril/valsartan may be less effective in AAs.

DETAILED DESCRIPTION:
To assess the efficacy and safety of sacubitril/valsartan in AA patients with HFrEF by comparing the outcomes of AA patients on ARNI therapy plus SOC (with or without hydralazine/isosorbide [H-IDSN]) to AA patients receiving ACEi/ARB therapy plus SOC (with or without H-ISDN).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as AA
* NYHA class II-IV symptoms
* Left ventricle EF <40%
* Receiving stable doses of standard therapy, including ACE inhibitors or ARBs, ARNI (within a month from discharge), combination H-ISDN, beta blockers, digoxin, spironolactone, and diuretics as tolerated.
* Patient must have minimum of three months follow-up

Exclusion Criteria:

* Patients not meeting inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: AAs with HFrEF on sacubitril/valsartan therapy
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Composite CV mortality or HF hospitalization | April 2017 to August 2020
  Composite CV mortality or HF hospitalization

SECONDARY OUTCOMES:
CV mortality | April 2017 to August 2020
  Individual components
HF hospitalization | April 2017 to August 2020
  Individual components
All-cause mortality | April 2017 to August 2020
  Individual components
New atrial fibrillation | April 2017 to August 2020
  Individual components
Renal function decline | April 2017 to August 2020
  Individual components
Change in EF | April 2017 to August 2020
  Individual components
Change in NYHA classification | April 2017 to August 2020
  Individual components

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Brown, PharmD, Principal Investigator — Methodist Dallas Medical Center Pharmacy
Locations (1):
- Methodist Dallas Medical Center Pharmacy, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided